CLINICAL TRIAL: NCT06998563
Title: The Effect of Lower Extremity Rotational Profile on Postural Control, Muscle Strength, Functional Capacity and Lower Extremity Function in Children With Generalized Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant Professor, Bezmialem Vakif University
Other Study IDs: 31.12.2024-177310
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Joint Hypermobility; Femoral Anteversion; Postural Control; Lower Extremity Muscle Strength; Functional Capacity; Lower Extremity Functional Scale; Rotational Malalignment of the Lower Extremity
Keywords: Generalized joint hypermobility; Lower extremity rotational profile; postural control; muscle strength; lower extremity functional scale; functional capacity
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Inclusion criteria for Group 1:
  Inclusion Criteria for Group 1:
  1. Being between 7-16 years old
  2. Having a body mass index within normal limits (18.5-24.9 kilogram/meter2)
  3. Beighton Score ≥ 5
  4. Having a lower extremity rotational profile problem according to Staheli rotational profile assessment
  Exclusion criteria for all groups;
  1. Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
  2. To have a surgical history associated with vertebral column and lower extremity
  3. Having cognitive, mental and/or serious psychiatric illness
  4. To participate in any exercise program or a sporty activity in the last six months
  Interventions: Other: Rotational Profile- Hip Internal and External Rotation Measurement; Other: Rotational Profile- Craig's Test Measurement; Other: Rotational Profile- Foot/Thigh Angle Measurement; Other: Rotational Profile- Heel Bisector Line Measurement; Other: Rotational Profile- Q Angle Measurement; Other: Rotational Profile- Navicular Drop Test Measurement; Other: Rotational Profile- Foot Progression Angle Measurement; Other: Muscle Shortness/Flexibility- Thomas Test Measurement; Other: Muscle Shortness/Flexibility- Popliteal Angle Measurement; Other: Muscle Shortness/Flexibility- Silfverskiöld Test Measurement; Other: Muscle Shortness/flexibility- Ober Test Measurement; Other: Muscle Shortnes/flexibility- Duncan-Ely Test Measurement; Other: Muscle Shortness/Flexibility- Sit-Reach Test Measurement; Other: Postural Control Assessment with Biodex Balance System (BBS); Other: Muscle Strength Assessment with Micro-FET2; Other: Functional Capacity Assessmnet with 6 Minute Walk Test Measurement; Other: Lower Extremity Functional Scale; Other: Pain Assessment with Viusal Analog Scale; Other: Demographic Information Form; Other: Ankle Joint Dorsiflexion Range of Motion Measurement; Other: Leg Length Measurement
- Group 2: Inclusion criteria for group 2:
  1. Being between 7-16 years old
  2. Having a body mass index within normal limits (18.5-24.9 kilogram/meter2)
  3. Beighton Score ≥ 5
  4. Having a normal lower extremity rotational profile problem according to Staheli rotational profile assessment
  Exclusion criteria for all groups;
  1. Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
  2. To have a surgical history associated with vertebral column and lower extremity
  3. Having cognitive, mental and/or serious psychiatric illness
  4. To participate in any exercise program or a sporty activity in the last six months
  Interventions: Other: Rotational Profile- Hip Internal and External Rotation Measurement; Other: Rotational Profile- Craig's Test Measurement; Other: Rotational Profile- Foot/Thigh Angle Measurement; Other: Rotational Profile- Heel Bisector Line Measurement; Other: Rotational Profile- Q Angle Measurement; Other: Rotational Profile- Navicular Drop Test Measurement; Other: Rotational Profile- Foot Progression Angle Measurement; Other: Muscle Shortness/Flexibility- Thomas Test Measurement; Other: Muscle Shortness/Flexibility- Popliteal Angle Measurement; Other: Muscle Shortness/Flexibility- Silfverskiöld Test Measurement; Other: Muscle Shortness/flexibility- Ober Test Measurement; Other: Muscle Shortnes/flexibility- Duncan-Ely Test Measurement; Other: Muscle Shortness/Flexibility- Sit-Reach Test Measurement; Other: Postural Control Assessment with Biodex Balance System (BBS); Other: Muscle Strength Assessment with Micro-FET2; Other: Functional Capacity Assessmnet with 6 Minute Walk Test Measurement; Other: Lower Extremity Functional Scale; Other: Pain Assessment with Viusal Analog Scale; Other: Demographic Information Form; Other: Ankle Joint Dorsiflexion Range of Motion Measurement; Other: Leg Length Measurement
- Control group: Criteria for inclusion for the control group;
  1. Being between 7-16 years
  2. Having body mass index at normal limits (18.5-24.9 kilogram/meter2)
  3. Beighton score <5
  4. Lower extremity rotational profile problem according to the steheli rotational profile evaluation is to be normal
  Exclusion criteria for all groups;
  1. To have any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
  2. To have a surgical history associated with vertebral column and lower extremity
  3. Having cognitive, mental and/or serious psychiatric illness
  4. To participate in any exercise program or a sporty activity in the last six months
  Interventions: Other: Rotational Profile- Hip Internal and External Rotation Measurement; Other: Rotational Profile- Craig's Test Measurement; Other: Rotational Profile- Foot/Thigh Angle Measurement; Other: Rotational Profile- Heel Bisector Line Measurement; Other: Rotational Profile- Q Angle Measurement; Other: Rotational Profile- Navicular Drop Test Measurement; Other: Rotational Profile- Foot Progression Angle Measurement; Other: Muscle Shortness/Flexibility- Thomas Test Measurement; Other: Muscle Shortness/Flexibility- Popliteal Angle Measurement; Other: Muscle Shortness/Flexibility- Silfverskiöld Test Measurement; Other: Muscle Shortness/flexibility- Ober Test Measurement; Other: Muscle Shortnes/flexibility- Duncan-Ely Test Measurement; Other: Muscle Shortness/Flexibility- Sit-Reach Test Measurement; Other: Postural Control Assessment with Biodex Balance System (BBS); Other: Muscle Strength Assessment with Micro-FET2; Other: Functional Capacity Assessmnet with 6 Minute Walk Test Measurement; Other: Lower Extremity Functional Scale; Other: Pain Assessment with Viusal Analog Scale; Other: Demographic Information Form; Other: Ankle Joint Dorsiflexion Range of Motion Measurement; Other: Leg Length Measurement

INTERVENTIONS:
Other: Rotational Profile- Hip Internal and External Rotation Measurement — Hip internal and external rotation angles measurement, hip range of motion evaluations will be performed. Measurements will be performed using a universal goniometer. The children will be positioned in the prone position with their knees flexed 90° and placed on the edge of the bed. The tuberositas tibia will be chosen as the pivot point of the goniometer, and the movable arm will be aligned with the tibial crista. The fixed arm will be placed perpendicular to the floor and the movable arm will be guided by the tibial crista. During hip rotation, it will be ensured that the hip remains stable and the movement occurs only in the hip joint.
  Other Names: Hip internal/external rotation measurement
Other: Rotational Profile- Craig's Test Measurement — The Craig's (Ryder) test, also known as the 'Trochanteric Prominence Angle Test', will be performed on the children included in the study according to the following protocol. The children will be placed in a prone position. The physiotherapist stood on the opposite side of the hip to be tested. The hips of the children will be placed in the extension position and the knee on the side to be tested will be held in the 90° flexion position. The physiotherapist palpated the trochanter major with the left hand and internal rotated the hip with the right hand. At the point where the trochanteric process will be most prominent, the angle between the tibia and the vertical plane will be measured using a goniometer and the femoral anteversion angle will be recorded.
  Other Names: Craig's test; Ryder test
Other: Rotational Profile- Foot/Thigh Angle Measurement — Foot/thigh angle assessment will be performed by measuring the angle between the long axis of the femur bone and the foot with a goniometer in the prone position. One arm of the goniometer will be placed parallel to the long axis of the femur, while the other arm will be placed so that it passes through the 2nd and 3rd metatarsals. Normally, the thigh-foot angle should be in external rotation between 10-15°. In young children, this angle can be considered normal up to 30°. A decrease in the thigh-foot angle will indicate internal tibial torsion (expressed as a negative value), which is the internal rotation of the tibia. In this case, there is an abnormal internal rotation of the tibia. If the measured foot-thigh angle exceeds 30°, it is considered to be external tibial torsion (external rotation of the tibia).
  Other Names: foot/thigh angle
Other: Rotational Profile- Heel Bisector Line Measurement — The heel bisector line test is an evaluation method that helps diagnose metatarsus adductus. During the test, the child will be placed in the prone position with the heel between the physiotherapist's fingers. Then, the midpoint of the lines drawn from the malleoli will be determined. From this point, a perpendicular line will be drawn from the heel to the toes along the foot axis with the help of a goniometer. Normally, this line should end between the 1st and 2nd toes. If the line ends at the 3rd, 4th or 5th toes, this may indicate the presence of metatarsus adductus.
  Other Names: heel bisector line
Other: Rotational Profile- Q Angle Measurement — The Q-angle is defined as the angle formed between an imaginary line connecting the anterior superior iliac spine of the pelvis to the midpoint of the patella and the proximal projection of the line from the tibial tubercle to the center of the patella. The child will first be placed in a supine position with legs extended and muscles relaxed, and the midpoint of the patella will be marked with a colored pencil. Then, the goniometer will be placed at the midpoint of the patella and care will be taken to fix the movable arm so that it points to the anterior superior iliac spine and the fixed arm so that it follows the tibia and the angle between the two will be recorded. The measurement will be recorded in two different positions, lying and standing. Q angle between 10-15° in boys and 15-20° in girls will be considered normal.
  Other Names: Q angle
Other: Rotational Profile- Navicular Drop Test Measurement — The navicular drop test is commonly used in clinics to assess pes planus. It will begin with the child sitting, feet flat on the floor, and no weight bearing. The navicular tubercle will be palpated and marked first, then the distance from the tubercle to the floor will be measured. The child will then stand with equal weight on both feet and the distance will be measured again. Measurements will be taken bilaterally and recorded in millimeters. The difference between the weighted and unweighted measurements will indicate foot posture: 5-9 millimeters is normal (neutral), 10 millimeters or more will indicate pronation (inward rotation), and 4 millimeters or less will indicate supination (outward rotation). This test is important for assessing the degree of pes planus.
  Other Names: navicular drop test
Other: Rotational Profile- Foot Progression Angle Measurement — The foot progression angle will be used as an important parameter in determining potential disorders and alignment errors in the child's walking pattern by reflecting the rotational relationships between the femur, tibia and foot. For this measurement, two chairs will first be placed opposite each other with a distance of 2 m between them. Then, the child will be asked to sit on the chair. In the sitting position, the middle of the heel and the second toe will be marked with colored paint. After the marking, the child will be asked to walk naturally on a flat surface to the chair opposite. The child will stand up from the sitting position and walk approximately 5-6 steps on a flat surface to the chair opposite. Then, the child will be asked to sit on the chair opposite and clean the paint off his foot. This colored marking will be made in a way that will create the child's walking traces. When the child finishes walking, these traces will be measured in degrees using a goniometer.
Other: Muscle Shortness/Flexibility- Thomas Test Measurement — The Thomas test will be performed to evaluate shortness/tightness in the hip flexor muscle group, especially in the iliopsoas muscle. The child will be placed in the supine position, the lumbar spine will be fixed and the assessment will begin. During the test, while the assessed hip is in knee extension, the opposite hip and knee will be passively flexed by the physiotherapist, and the hip movement of the assessed side will be observed during this time. The Thomas test will be recorded as negative if no flexion movement is observed in the assessed hip. In the presence of shortness/tightness, the assessed hip is seen to be flexed, and in this case, the Thomas test will be recorded as positive.
  Other Names: thomas test
Other: Muscle Shortness/Flexibility- Popliteal Angle Measurement — The popliteal angle test will be used to evaluate shortness or tightness of the hamstring muscles. The hip and knee will be placed in a 90° flexion position while the child is in the supine position. While the physiotherapist passively moves the knee joint towards extension, the popliteal angle will be measured using a goniometer. While one arm of the goniometer is placed parallel to the lateral surface of the femur, the other arm is held parallel to the fibula head and the angle will be measured. The knee joint will be extended until it encounters resistance and the angle between the tibia and the vertical plane will be recorded as the popliteal angle.
  Other Names: popliteal angle
Other: Muscle Shortness/Flexibility- Silfverskiöld Test Measurement — Gastrocnemius assessment will be evaluated with the Silfverskiold test for all children participating in the study. The assessment will be performed bilaterally in supine positions where the child does not bear weight on their feet. The knee joint will be in full extension and 90° flexion, the subtalar joint will be in a neutral position, and the ankle dorsiflexion will be measured with the fixed arm of the universal goniometer on the fibula shaft and the mobile arm following the fifth metatarsal shaft. The measured angles will be recorded in degrees (°). Passive ankle dorsiflexion of ≤ 10° with the knee extended and a minimum of 10° increase in dorsiflexion with the knee flexed will be considered as isolated gastrocnemius muscle shortness.
  Other Names: silfverskiöld test
Other: Muscle Shortness/flexibility- Ober Test Measurement — The Ober test will be performed to measure the length of the iliotibial band. Both the Ober test and the modified Ober test are widely used and accepted tests to assess iliotibial band length. During the test, the child will be placed in a supine position with the lower leg slightly bent at the hip and knee. The upper leg will be in 90° flexion of the knee. Once positioning is complete, the physiotherapist will hold the ankle of the upper leg with one hand and stabilize the hip with the other hand. The leg will then be abducted and the knee extended and the leg moved until the femur is in line with the body. Finally, the thigh will be allowed to fall towards the surface in this plane and the result of the test will be judged by the amount of adduction of the hip. If the knee hangs in the air, the test is positive. If the knee falls, the test is negative
  Other Names: ober test
Other: Muscle Shortnes/flexibility- Duncan-Ely Test Measurement — The Duncan-Ely test will be used to evaluate the shortness and tightness of the rectus femoris muscle. While the child is lying in the prone position, the hip will be fixed with one hand by the physiotherapist and the hip and knee will be kept in extension. In this position, the knee joint will be passively flexed in order to stretch the rectus femoris muscle on the tested side. If no shortness or tightness is observed in the rectus femoris muscle on the same side during the test and hip extension is maintained, the Duncan-Ely test will be recorded as negative. However, when the knee is flexed and a flexion movement is observed in the hip, the test will be recorded as positive.
  Other Names: duncan-ely test
Other: Muscle Shortness/Flexibility- Sit-Reach Test Measurement — The Sit-Reach test will be used to evaluate the flexibility of the hamstring and lower back muscle groups. The S&R Sit and Reach® table will be used for this test. The child will sit in front of the table with dimensions of 55 centimeters long, 35 centimeters wide, and 30 centimeters high, and his/her feet will be positioned on the foot surface of the table. The child will be asked to place his/her hands on top of each other and stretch forward in a slow and controlled manner, bringing the ruler on the table forward. He/she will be asked to wait 1-2 seconds at the farthest point without stretching forward or backward. Scoring will be done according to the ruler on the table. (On this table, the child's ability to bring the ruler to the tips of his/her toes corresponds to 23 centimeters). The test will be repeated three times for each child to ensure reliability, and the highest value will be recorded in centimeters.
  Other Names: sit-reach test
Other: Postural Control Assessment with Biodex Balance System (BBS) — Postural stability, limits of stability, and sensory integration of balance will be assessed using the Biodex Balance System®. Biodex Balance System is a validated and reliable device used to evaluate postural stability, limits of stability, and fall risk. It consists of a balance platform, arm supports, a screen, and a printer. The platform can be set to static or dynamic mode (12 levels; level 12 = most stable, level 1 = least stable with up to 20° movement in all directions). Prior to testing, children will be informed about the procedures. The heel and toe positions will be recorded based on medial-lateral (B-J), anterior, and posterior (1-21) axes. Arm support and screen height will be individually adjusted. Child-specific posture and identification data will be entered into the system. Three tests will be performed: postural stability, limits of stability, and sensory integration of balance.
  Other Names: Biodex Balance System
Other: Muscle Strength Assessment with Micro-FET2 — Muscle tests will be performed using the MicroFET 2 digital hand dynamometer according to the device manual. The measurement will be performed in supine, prone, side-lying and sitting positions by preventing compensatory movements. During the test, the arms will be positioned so that they will not receive power from anywhere on/to the side of the body. Measurements will be performed bilaterally. While the child to whom the test is applied is expected to perform the requested movement with all his/her strength, the evaluating physiotherapist will apply resistance in the opposite direction in proportion to the strength. During the evaluation of the same muscle, a 30-second break will be given between repetitions, and a five-minute rest will be given before moving on to the test for a different muscle. Isometric muscle strength of the Iliopsoas, Gluteus Maximus, Gluteus Medius, Quadriceps, Hamstring, Tibialis Anterior, and Gastrosoleus muscles will be evaluated.
  Other Names: Micro-FET2
Other: Functional Capacity Assessmnet with 6 Minute Walk Test Measurement — The 6MWT will be done on a flat 30-meter track marked every 3 meters, with clear start and finish lines. Before the test, the child rests 15 minutes while contraindications will be checked. If none, blood pressure, oxygen saturation, pulse, and Borg scale scores for dyspnea and fatigue will be recorded. Medications taken will be noted. The child will be instructed to walk at their own pace for 6 minutes, allowed to stop or rest, and continue until "test is over" is announced. The test will start with "test is started" and end with "test is over." The timer will run continuously even if paused. The test ends if chest pain, severe breathlessness, cramps, unsteadiness, sweating, pallor, or oxygen saturation <85% occurs. Afterward, the child will be sits and post-test vitals and Borg scores will be recorded. Distance walked and any complaints during the test will be noted.
  Other Names: 6MWT
Other: Lower Extremity Functional Scale — The Lower Extremity Functional Scale will be used to evaluate the functional ability of the entire lower extremity in individuals with musculoskeletal disorders. This scale will question the difficulty experienced in various daily activities due to the problem in the lower extremity with 20 items. Each item will be scored between 0-4 on a Likert scale (0=extremely difficult/too difficult to do the activity; 4=not difficult at all). The total score varies between 0-80 and the higher the score, the higher the functional level. A validity and reliability study has been conducted for the Turkish version of the scale to be used in evaluating lower extremity functions.
  Other Names: LEFS
Other: Pain Assessment with Viusal Analog Scale — The Visual Analog Scale is a simple and reliable tool that is widely used to assess subjective experiences such as pain. It consists of a 10 cm horizontal line with one end indicating "no pain" and the other end indicating "worst pain imaginable". Individuals will mark the point that reflects their perception of intensity, which will then be measured in millimeters or centimeters to obtain a numerical score. Higher values will indicate greater severity. The Visual Analog scale is valid and reliable in a variety of populations and conditions, including musculoskeletal pain.
  Other Names: VAS
Other: Demographic Information Form — All children's gender, age, body weight, height and dominant side information will be recorded before clinical evaluations. The body mass index (kilogram/meter2) of the child will be calculated and recorded with the recorded body weight (kilogram) and height (meter) values.
Other: Ankle Joint Dorsiflexion Range of Motion Measurement — Dorsiflexion range of motion with the knee joint in full extension and 90° flexion, the subtalar joint in a neutral position, the ankle dorsiflexion will be measured with the fixed arm of the universal goniometer on the fibula shaft and the mobile arm following the fifth metatarsal shaft. The measured angles were recorded in degrees (°). Measurements will be made bilaterally.
  Other Names: ROM
Other: Leg Length Measurement — Leg Length Measurement, the child will be placed in a supine position. The legs will be positioned in extension and the muscles will be relaxed. The physiotherapist will measure and record the child's right leg length from the SIAS bone to the medial malleola with a flexible metal tape measure. Measurements will be made bilaterally.

SUMMARY:
Generalized joint hypermobility is when the range of motion in synovial joints exceeds its physiological limits. The aim of this investigation is to investigate the effect of lower extremity rotational profile on postural control, muscle strength, functional capacity and lower extremity function in children with generalized joint hypermobility. Within the scope of this cross-sectional study, permission was obtained from Bezmialem Vakif University Non-Interventional Clinical Research Ethics Committee with the decision number 177310 dated 31.12.2024. Following the Ethics Committee approval, data collection started and the study will be conducted in accordance with the Declaration of Helsinki. "Informed Voluntary Consent Form" prepared for both parents and children and approved by Bezmialem Vakıf University Non-Interventional Clinical Research Ethics Committee will be signed.

All children participating in the study and their parents will be informed about the study and those who voluntarily agree to participate in the study will be invited by appointment.

All evaluations will be carried out in the Pediatric and Cardiac Physiotherapy and Rehabilitation Education and Research Laboratories of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Bezmialem Vakıf University. Forty-eight children who meet the specified inclusion/exclusion criteria will be included in the study sample.

Within the scope of the study, demographic information of the children will be recorded with the sociodemographic evaluation form and clinical evaluations will be performed on the same day. All assessments will be administered to all children in all three groups by the same researcher in the following order.

The evaluation process will start with the completion of the sociodemographic information form. Then, the general joint hypermobility status of the participants will be evaluated with the Beighton Score. Within the scope of clinical measurements, bilateral lower extremity rotational profile will be determined by Craig's test, foot-thigh angle, foot progression angle, navicular drop test, Heel Bisector Line Test and Q angle measurements. Lower extremity muscle shortness and flexibility will be evaluated using bilateral Thomas test, Duncan-Ely test, Ober test, popliteal angle test, Silfverskiöld test and sit-to-stand test. Bilateral hip internal and external rotation angles and ankle dorsiflexion angle measurements will be performed to measure range of motion. Bilateral leg length measurements will be performed and general pain status will be questioned using the Visual Analog Scale.

Postural control will be assessed using the Biodex Balance System, muscle strength will be assessed using the MicroFET2 hand dynamometer, functional capacity will be assessed using the 6-minute walk test and lower extremity functionality will be assessed using the Lower Extremity Functional Scale .

DETAILED DESCRIPTION:
Generalized joint hypermobility is characterized by an excessive range of motion in multiple joints without the presence of hereditary connective tissue disorders. Despite the clinical relevance of biomechanical changes such as increased femoral anteversion in children with Generalized Joint Hypermobility , limited research exists on how these alterations affect postural control, muscle strength, functional capacity, and lower extremity function. This observational cross-sectional study aims to evaluate the influence of lower extremity rotational profile on these parameters in children with Generalized Joint Hypermobility.

The sample size of the study was calculated with G*Power 3.1.9.4 analysis program. In the calculation of the sample size, 6-minute walking distance, one of the parameters evaluated in the study of Kepenek-Varol et al. in which individuals with generalized joint hypermobility were compared with their healthy peers, was taken into consideration. The analysis was performed with a priori power analysis ANOVA (one-way) approach for three groups. Accordingly, while the effect size obtained was Cohen's d = 0.64, the total minimum sample size to be reached for the three groups was calculated as 42 individuals in order to obtain 95% power at α=0.05 level. Considering that there may be missing data during the research phase, this number was increased by 10% and the number of participants for each group was determined as 16 and 48 people in total. This study will include a total of 48 children who will be divided into three groups.

Inclusion Criteria for Group 1:

1. Being between 7-16 years old
2. Having a body mass index within normal limits (18.5-24.9 kilograms/meter2)
3. Beighton Score ≥ 5
4. Having a lower extremity rotational profile problem according to Staheli rotational profile assessment

Inclusion Criteria for Group 2:

1. Being between 7-16 years old
2. Having a body mass index within normal limits (18.5-24.9 kilograms/meter2)
3. Beighton Score ≥ 5
4. Having a normal lower extremity rotational profile problem according to Staheli rotational profile assessment

Inclusion Criteria for the Control Group;

1. Being between 7-16 years old
2. Having a body mass index within normal limits (18.5-24.9 kilograms/meter2)
3. Beighton Score < 5
4. Having a normal lower extremity rotational profile problem according to Staheli rotational profile assessment

Exclusion criteria for all groups;

1. Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
2. History of surgery related to the vertebral column and lower extremities
3. Having cognitive, mental and/or severe psychiatric illness
4. Participated in any exercise program or sportive activity in the last six months

Applications will be carried out in the Cardiac Physiotherapy and Rehabilitation Education and Research Laboratories of Bezmialem Vakif University Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation after permission is obtained.

Within the scope of this cross-sectional study, permission was obtained from Bezmialem Vakif University Non-Interventional Clinical Research Ethics Committee with the decision number 177310 dated 31.12.2024. Following the approval of the Ethics Committee, data collection will begin and the study will be conducted in accordance with the Declaration of Helsinki. "Informed Voluntary Consent Form" prepared for both parents and children and approved by Bezmialem Vakıf University Non-Interventional Clinical Research Ethics Committee will be signed.

All children participating in the study and their parents will be informed about the study and those who voluntarily agree to participate in the study will be invited by appointment.

All evaluations will be performed in the Pediatric and Cardiac Physiotherapy and Rehabilitation Education and Research Laboratories of the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Bezmialem Vakif University. Forty-eight children who meet the specified inclusion/exclusion criteria will be included in the study sample.

Within the scope of the study, demographic information of the children will be recorded with the sociodemographic evaluation form and clinical evaluations will be performed on the same day. All assessments will be administered to all children in all three groups by the same researcher in the following order.

The evaluation process will start with the completion of the sociodemographic information form. Then, the general joint hypermobility status of the participants will be evaluated with the Beighton Score. Within the scope of clinical measurements, bilateral lower extremity rotational profile will be determined by hip internal and external rotation measurements, Craig's test, foot-thigh angle, heel bisector line, Q angle, navicular drop test and foot progression angle. Lower extremity muscle shortness and flexibility will be evaluated using bilateral Thomas test, popliteal angle test, Silfverskiöld test, Ober test, Duncan-Ely and sit-to-stand test. Bilateral ankle dorsiflexion angle and bilateral leg length measurements will be performed to measure range of motion. General pain status will be questioned using the Visual Analog Scale.

Postural control will be assessed with the Biodex Balance System, muscle strength with the MicroFET2 hand dynamometer, functional capacity with the 6-minute walk test and lower extremity functionality with the Lower Extremity Functional Scale.

In order to prevent fatigue from having a negative effect on the test results, the order of administration of each test will be determined in accordance with the position of the children. Lying tests will be performed in the supine position, while prone tests will be performed in the prone position. Standing tests will be performed in the standing position respectively. During the assessments, children will be tested in their underwear only and the temperature of the environment will be controlled to ensure their comfort. Only researchers and children will be present in the laboratory to avoid distractions during the tests.

Demographic information form All children's gender, age, body weight, height and dominant side information will be recorded before clinical evaluations. The body mass index (kilogram/meter2) of the child will be calculated and recorded with the recorded body weight (kilogram) and height (meter) values.

Clinical evaluations:

Evaluation of joint hypermobility according to the Beighton score:

The Beighton Score is one of the most preferred scoring methods due to its bilateral evaluation of the joints and easy applicability. It was created by Beighton in 1973 by modifying the Carter and Wilkinson criteria. The Beighton Score is a valid and reliable measurement tool that is widely used in the evaluation of joint hypermobility in childhood and adolescence. In this study, the Beighton Score will be used to define asymptomatic generalized joint hypermobility. Although variable threshold values have been proposed in the literature according to different age groups, in this study, a Beighton score of ≥5 points and above will be accepted as the criterion for hypermobility in children aged 7-16 years. Children who reach this threshold are classified as children with generalized joint hypermobility.

The Beighton Score is a measurement tool evaluated over a total of 9 points. The evaluation is based on the following criteria:

* Passive dorsiflexion of the 5th finger in both hands exceeding 90° (1 point per side),
* Contact of the thumb with the volar side (flexor side) of the forearm with flexion in both hands (1 point per side),
* Hyperextension of more than 10° at both elbows (1 point per side),
* Hyperextension of more than 10° in both knees (1 point per side),
* Palms touching the ground during forward flexion of the trunk with the knees in extension (1 point).

Evaluation of lower limb rotational profile:

In the study, Staheli's rotational profile tests will be applied to evaluate the rotational profile of the lower extremities of the children. All children in all three groups underwent the following tests;

Hip internal and external rotation angles measurement:

In the study, hip range of motion evaluations will be performed. Measurements will be performed using a universal goniometer. The children will be positioned in the prone position with their knees flexed 90° and placed on the edge of the bed. The tuberositas tibia will be chosen as the pivot point of the goniometer, and the movable arm will be aligned with the tibial crista. The fixed arm will be placed perpendicular to the floor and the movable arm will be guided by the tibial crista. During hip rotation, it will be ensured that the hip remains stable and the movement occurs only in the hip joint.

Craig's test The Ryder test, also known as the 'Trochanteric Prominence Angle Test', will be performed on the children included in the study according to the following protocol. The children will be placed in a prone position. The physiotherapist stood on the opposite side of the hip to be tested. The hips of the children will be placed in the extension position and the knee on the side to be tested will be held in the 90° flexion position. The physiotherapist palpated the trochanter major with the left hand and internal rotated the hip with the right hand. At the point where the trochanteric process will be most prominent, the angle between the tibia and the vertical plane will be measured using a goniometer and the femoral anteversion angle will be recorded.

Foot/thigh angle measurement:

This assessment will be performed by measuring the angle between the long axis of the femur bone and the foot with a goniometer in the prone position. One arm of the goniometer will be placed parallel to the long axis of the femur, while the other arm will be placed so that it passes through the 2nd and 3rd metatarsals. Normally, the thigh-foot angle should be in external rotation between 10-15°. In young children, this angle can be considered normal up to 30°. A decrease in the thigh-foot angle will indicate internal tibial torsion (expressed as a negative value), which is the internal rotation of the tibia. In this case, there is an abnormal internal rotation of the tibia. If the measured foot-thigh angle exceeds 30°, it is considered to be external tibial torsion (external rotation of the tibia).

Heel bisector line:

The heel bisector line test will be an evaluation method that helps diagnose metatarsus adductus. During the test, the child will be placed in the prone position with the heel between the physiotherapist's fingers. Then, the midpoint of the lines drawn from the malleoli will be determined. From this point, a perpendicular line will be drawn from the heel to the toes along the foot axis with the help of a goniometer. Normally, this line should end between the 1st and 2nd toes. If the line ends at the 3rd, 4th or 5th toes, this may indicate the presence of metatarsus adductus.

Q angle measurement:

Q-angle is defined as the angle formed between an imaginary line connecting the anterior superior iliac spine of the pelvis to the midpoint of the patella and the proximal projection of the line extending from the tibial tubercle to the center of the patella. The child will first be placed in a supine position, with legs extended and muscles relaxed, and the midpoint of the patella is marked with a colored pencil. Then, the goniometer will be placed at the exact midpoint of the patella, and care is taken to fix the mobile arm so that it points to the anterior superior iliac spine and the fixed arm so that it follows the tibia, and the angle in between will be recorded. The measurement will be recorded in two different positions: lying down and standing. The Q angle is considered normal between 10-15 ° in boys and 15- 20 ° in girls.

Navicular drop test:

The navicular drop test is a widely used test in the clinic to evaluate the presence and degree of pes planus. This test will be started with the child in a sitting position, with the feet only in contact with the floor, without weight bearing. In the first step, the navicular tubercle will be palpated and marked. While the child is in a sitting position, the distance between the navicular tubercle and the floor will be measured. This measurement will be made when the feet are only in contact with the floor without any weight bearing. Then, the child is asked to stand and the distance between the navicular tubercle and the floor will be measured again in a position where the feet are equally weight bearing. Measurements will be made bilaterally, separately for each foot, and the results will be recorded in millimeters.

In the navicular drop test, the difference between weighted and unweighted measurements is interpreted as follows: Differences between 5-9 millimeter are considered normal (neutral), differences of 10 milimeter and above are considered as an indicator of pronation (inward rotation) in the foot, while differences of 4 millimeter and below are associated with supination (outward rotation) in the foot. This test is an important measurement tool for determining the degree of pes planus

Foot progression angle:

Foot progression angle is used as an important parameter in determining potential disorders and alignment errors in the child's walking pattern by reflecting the rotational relationships between the femur, tibia and foot. For this measurement, two chairs will first be placed opposite each other with a distance of 2 m between them. Then, the child will be asked to sit on the chair. In the sitting position, the middle of the heel and the second toe will be marked with colored paint. After the marking, the child will be asked to walk naturally on a flat surface to the chair opposite. The child will stand up from the sitting position and walk approximately 5-6 steps on a flat surface to the chair opposite. Then, the child will be asked to sit on the chair opposite and clean the paint on his foot. This colored marking will be made in a way that will create the child's walking traces. When the child finishes walking, these traces will be measured in degrees using a goniometer. To measure the foot progression angle with a goniometer; One arm will be positioned so that it is aligned with the direction of the footprints, and the other arm will be positioned parallel to the axis of the tibia. The angle between the foot and the tibia will be recorded in degrees with a goniometer.

Measurement of ankle joint dorsiflexion range of motion:

With the knee joint in full extension and 90° flexion, the subtalar joint in a neutral position, the ankle dorsiflexion will be measured with the fixed arm of the universal goniometer on the fibula shaft and the mobile arm following the fifth metatarsal shaft. The measured angles will be recorded in degrees (°). Measurements will be made bilaterally.

Leg length measurement:

The child will be placed in a supine position. The legs will be positioned in extension and the muscles will be relaxed. The physiotherapist will measure and record the child's right leg length from the anterior superior iliac spine bone to the medial malleolus with a flexible metal tape measure. Measurements will be made bilaterally.

Muscle shortness/flexibility assessments

Thomas test:

The Thomas test will be performed to evaluate shortness/tightness in the hip flexor muscle group, especially in the iliopsoas muscle. The child will be placed in the supine position, the lumbar spine will be fixed and the assessment will begin. During the test, while the assessed hip is in knee extension, the opposite hip and knee will be passively flexed by the physiotherapist, and the hip movement of the assessed side will be observed during this time. The Thomas test will be recorded as negative if no flexion movement is observed in the assessed hip. In the presence of shortness/tightness, the assessed hip is seen to be flexed, and in this case, the Thomas test will be recorded as positive.

Popliteal angle test:

The popliteal angle test will be used to evaluate shortness or tightness of the hamstring muscles. The hip and knee will be placed in a 90° flexion position while the child is in the supine position. While the physiotherapist passively moves the knee joint towards extension, the popliteal angle will be measured using a goniometer. While one arm of the goniometer is placed parallel to the lateral surface of the femur, the other arm is held parallel to the fibula head and the angle will be measured. The knee joint will be extended until it encounters resistance and the angle between the tibia and the vertical plane will be recorded as the popliteal angle.

Silfverskiold test:

Gastrocnemius assessment will be evaluated with the Silfverskiold test for all children participating in the study. The assessment will be performed bilaterally in supine positions where the child does not bear weight on their feet. The knee joint will be in full extension and 90° flexion, the subtalar joint will be in a neutral position, and the ankle dorsiflexion will be measured with the fixed arm of the universal goniometer on the fibula shaft and the mobile arm following the fifth metatarsal shaft. The measured angles will be recorded in degrees (°). Passive ankle dorsiflexion of ≤ 10° with the knee extended and a minimum of 10° increase in dorsiflexion with the knee flexed will be considered as isolated gastrocnemius muscle shortness.

Ober test:

The Ober test will be an assessment performed to measure the length of the iliotibial band. There are also some modifications of this test, such as the modified Ober test described by Kendall in 1953. Both the Ober test and the modified Ober test are widely used and accepted tests to assess iliotibial band length. During the test, the child will be placed in a side-lying position with the lower leg slightly flexed at the hip and knee. The knee of the upper leg is ensured to be in 90° flexion. After the positioning is completed, the physiotherapist will hold the ankle of the upper leg with one hand and stabilize the hip with the other hand. Then, the leg will be abducted and the knee will be extended, and the leg will be moved until the femur is in line with the body. Finally, the thigh will be allowed to fall towards the surface in this plane, and the result of the test will be evaluated according to the amount of adduction of the hip. If the knee hangs in the air, the test will be recorded as positive. If the leg falls towards the surface, the test will be evaluated as negative.

Duncan-ely test:

The Duncan-Ely test will be used to evaluate the shortness and tightness of the rectus femoris muscle. While the child is lying in the prone position, the hip will be fixed with one hand by the physiotherapist and the hip and knee will be kept in extension. In this position, the knee joint will be passively flexed in order to stretch the rectus femoris muscle on the tested side. If no shortness or tightness is observed in the rectus femoris muscle on the same side during the test and hip extension is maintained, the Duncan-Ely test will be recorded as negative. However, when the knee is flexed and a flexion movement is observed in the hip, the test will be recorded as positive.

Sit-reach test:

This test is a frequently used test to evaluate the flexibility of the hamstring and lower back muscle groups. The S&R Sit and Reach® table will be used for this test. The child will sit in front of the table with dimensions of 55 centimeters long, 35 centimeters wide, and 30 centimeters high, and his/her feet will be positioned on the foot surface of the table. The child will be asked to place his/her hands on top of each other and stretch forward in a slow and controlled manner, bringing the ruler on the table forward. He/she will be asked to wait 1-2 seconds at the farthest point without stretching forward or backward. Scoring will be done according to the ruler on the table. (On this table, the child's ability to bring the ruler to the tips of his/her toes corresponds to 23 centimeters). The test will be repeated three times for each child to ensure reliability, and the highest value will be recorded in centimeters.

Postural control assessment with Biodex balance system Biodex Balance System is a valid and reliable equipment that will be used to assess postural stability, stability limits and fall risk. It consists of a balance platform, arm supports, a screen and printer. The platform can be adjusted as static or mobile (12 levels of movement amount; level 12 is the most stable, level 1 is the least stable level that can move up to 20 degrees in each direction) according to the test that will be applied. Before the evaluation, explanatory information about the test steps will be given to all children included in the study. The axes where the heel and toe tips of each child will be recorded according to the medial and lateral (B, C, D, E, F, G, H, I, J) axes, the angles in the anterior and the axes in the posterior (1, 2, 3…,21). The arm support and test screen height will be adjusted specifically for each child. The child's information and stance position information will be entered into the balance beam screen. The device will be evaluated with three separate tests: postural stability test, stability limits test and balance sensory integration test.

Postural Stability (Test of Postural Stability) This test will evaluate the child's ability to maintain the center of balance on a stable platform and record the deviations from the center. General, anterior/posterior and medial/lateral stability indexes will be calculated and recorded as degrees. The general stability index reflects the variability of the platform relative to the horizontal plane during all movements performed in the test. Anterior/posterior stability index reflects the variability for movements in the sagittal plane, medial/lateral stability index reflects the variability for movements in the frontal plane. A high score value will indicate that postural stability is affected more. In this test, three 20-second measurements will be made with 10 seconds between each measurement.

Stability limits test This test, performed on a static platform, will evaluate the child's ability to move and control the center of gravity between the body's support surfaces. Directional control (general, forward, backward, left, right, forward/left, forward/right, backward/left, backward/right) will be evaluated and expressed as a percentage value. High scores indicate good postural control (100% = perfect control).

Sensory integration of balance test This test will evaluate how the child's various senses contribute to balance and how well they can compensate for balance when one or more of these senses are eliminated. The test will be performed on a hard surface with the static platform setting, with eyes open, eyes closed, and on a foam surface with eyes open, eyes closed, and the sway index values will be recorded for each of the four positions. In this test, four measurements will be made with a 10-second rest between each measurement and each test duration of 30 seconds.

Lower extremity muscle strength measurement Micro-FET2:

Muscle tests will be performed using the MicroFET 2 digital hand dynamometer according to the device manual. The measurement will be performed in supine, prone, side-lying and sitting positions by preventing compensatory movements. During the test, the arms will be positioned so that they will not receive power from anywhere on/to the side of the body. Measurements will be performed bilaterally. While the child to whom the test will be applied is expected to perform the requested movement with all his/her strength, the evaluating physiotherapist will apply resistance in the opposite direction in proportion to the strength. During the evaluation of the same muscle, a 30-second break will be given between repetitions, and a five-minute rest will be given before moving on to the test for a different muscle. Isometric muscle strength of the Iliopsoas, Gluteus Maximus, Gluteus Medius, Quadriceps, Hamstring, Tibialis Anterior, and Gastrosoleus muscles will be evaluated in the measurement. Strength measurements will be repeated 3 times and the highest measured strength value will be recorded with a kilogram/force value and evaluated.

6-Minute Walking test: The test will be performed on a smooth and flat track that is 30 meters long, marked every 3 meters, and the start and finish lines are marked with a visible line. Before starting the test, the child will rest in a chair for 15 minutes. During this time, the patient's contraindications for the 6-minute walking test will be questioned. If there are no contraindications, the patient's blood pressure, oxygen saturation with a pulse oximeter, pulse, and the patient's dyspnea and fatigue level according to the Borg scale will be checked after the patient rests. If any medications are taken before the test, these will be recorded. The child will be brought to the starting line. The child will be given; The patient is informed that the patient should walk at their own pace for 6 minutes on the track, that they can end the test at any time if they have any complaints, that they can stop and rest if needed during the test and that they should continue the test until the command "test is over" is given, and the chronometer is started and the test will be started with the command "test is started" and the test will be ended with the command "test is over". If the patient stops and rests during the test and pauses the test, the chronometer will not be stopped. The test will be ended if the child has chest pain, intolerable shortness of breath, leg cramps, staggering, diaphoresis, bruising or pallor and oxygen saturation is <85%. After the test is over, the child is seated on a chair, the patient's oxygen saturation, pulse and dyspnea and fatigue levels according to the Borg scale will be checked with a pulse oximeter and the distance the patient walked for 6 minutes will be calculated and the test will be ended. If the child has complaints such as chest pain, dizziness, hip pain or leg pain during the test, it will be recorded.

Lower extremity functional scale:

The Lower Extremity Functional Scale is a questionnaire that will be used to evaluate the functional ability of the entire lower extremity in individuals with musculoskeletal disorders. This scale will question the difficulty experienced in various daily activities due to the problem in the lower extremity with 20 items. Each item is scored between 0-4 on a Likert scale (0=extremely difficult/too difficult to do the activity; 4=not difficult at all). The total score varies between 0-80 and the higher the score, the higher the functional level. A validity and reliability study has been conducted for the Turkish version of the scale to be used in evaluating lower extremity functions.

The Statistical Package for the Social Sciences 26.0 for Windows package program will be used in the statistical analysis of the data obtained. Descriptive statistics (mean±standard deviation, minimum-maximum, number and percentile) will be given for discrete and continuous variables. Groups will be compared with one-way ANOVA. Post hoc test will be performed according to normality with the Shapiro-Wilk test and homogeneity of variance between groups with Levene's test. Categorical groups will be compared with the chi-square (χ2) test. p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria for Group 1:

1. Being between 7-16 years old
2. Having a body mass index (BMI) within normal limits (18.5-24.9 kg/m2)
3. Beighton Score ≥ 5
4. Having a lower extremity rotational profile problem according to Staheli rotational profile assessment

Inclusion Criteria for Group 2:

1. Being between 7-16 years old
2. Having a BMI within normal limits (18.5-24.9 kg/m2)
3. Beighton Score ≥ 5
4. Having a normal lower extremity rotational profile problem according to Staheli rotational profile assessment

Inclusion Criteria for the Control Group;

1. Being between 7-16 years old
2. Having a BMI within normal limits (18.5-24.9 kg/m2)
3. Beighton Score < 5
4. Having a normal lower extremity rotational profile problem according to Staheli rotational profile assessment

Exclusion criteria for all groups;

1. Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
2. History of surgery related to the vertebral column and lower extremities
3. Having cognitive, mental and/or severe psychiatric illness
4. Participated in any exercise program or sportive activity in the last six months

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Study Population: The sample size of the study was calculated with the G*Power 3.1.9.4 analysis program. In the calculation of the sample size, 6-minute walking distance, one of the parameters evaluated in the study of Kepenek-Varol et al. in which individuals with generalized joint hypermobility were compared with their healthy peers, was taken into consideration. The analysis was performed with a priori power analysis ANOVA (One-way) approach for the three groups. Accordingly, the effect size obtained was Cohen's d = 0.64, while the total minimum sample size to be reached for the three groups was calculated as 42 individuals in order to obtain 95% power at α=0.05 level. Considering that there might be missing data during the research phase, this number was increased by 10% and the number of participants for each group was determined as 16 and 48 in total.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-12 (Actual)

PRIMARY OUTCOMES:
Rotational Profile- Hip Internal and External Rotation Measurement | Day 1
  Hip internal and external rotation angles measurement, hip range of motion evaluations will be performed. Measurements will be performed using a universal goniometer. The children will be positioned in the prone position with their knees flexed 90° and placed on the edge of the bed. The tuberositas tibia will be chosen as the pivot point of the goniometer, and the movable arm will be aligned with the tibial crista. The fixed arm will be placed perpendicular to the floor and the movable arm will be guided by the tibial crista. During hip rotation, it will be ensured that the hip remains stable and the movement occurs only in the hip joint.
Rotational Profile- Craig's Test Measurement | Day 1
  The Craig's (Ryder) test, also known as the 'Trochanteric Prominence Angle Test', will be performed on the children included in the study according to the following protocol. The children will be placed in a prone position. The physiotherapist stood on the opposite side of the hip to be tested. The hips of the children will be placed in the extension position and the knee on the side to be tested will be held in the 90° flexion position. The physiotherapist palpated the trochanter major with the left hand and internal rotated the hip with the right hand. At the point where the trochanteric process will be most prominent, the angle between the tibia and the vertical plane will be measured using a goniometer and the femoral anteversion angle will be recorded.
Rotational Profile- Foot/Thigh Angle Measurement | Day 1
  Foot/thigh angle, assessment will be performed by measuring the angle between the long axis of the femur bone and the foot with a goniometer in the prone position. One arm of the goniometer will be placed parallel to the long axis of the femur, while the other arm will be placed so that it passes through the 2nd and 3rd metatarsals. Normally, the thigh-foot angle should be in external rotation between 10-15°. In young children, this angle can be considered normal up to 30°. A decrease in the thigh-foot angle will indicate internal tibial torsion (expressed as a negative value), which is the internal rotation of the tibia. In this case, there is an abnormal internal rotation of the tibia. If the measured foot-thigh angle exceeds 30°, it is considered to be external tibial torsion (external rotation of the tibia).
Rotational Profile- Heel Bisector Line Measurement | Day 1
  The heel bisector line test is an evaluation method that helps diagnose metatarsus adductus. During the test, the child will be placed in the prone position with the heel between the physiotherapist's fingers. Then, the midpoint of the lines drawn from the malleoli will be determined. From this point, a perpendicular line will be drawn from the heel to the toes along the foot axis with the help of a goniometer. Normally, this line should end between the 1st and 2nd toes. If the line ends at the 3rd, 4th or 5th toes, this may indicate the presence of metatarsus adductus.
Rotational Profile- Q Angle Measurement | Day 1
  Q-angle is defined as the angle formed between an imaginary line connecting the anterior superior iliac spine of the pelvis to the midpoint of the patella and the proximal projection of the line extending from the tibial tubercle to the center of the patella. The child will first be placed in a supine position, with legs extended and muscles relaxed, and the midpoint of the patella will be marked with a colored pencil. Then, the goniometer will be placed at the exact midpoint of the patella, and care is taken to fix the mobile arm so that it points to the anterior superior iliac spine and the fixed arm so that it follows the tibia, and the angle in between will be recorded. The measurement will be recorded in two different positions: lying down and standing. The Q angle is considered normal between 10-15 ° in boys and 15- 20 ° in girls.
Rotational Profile- Navicular Drop Test Measurement | Day 1
  The navicular drop test is commonly used in clinics to assess pes planus. It will begin with the child sitting, feet flat on the floor, and no weight bearing. The navicular tubercle will be palpated and marked first, then the distance from the tubercle to the floor will be measured. The child will then stand with equal weight on both feet and the distance will be measured again. Measurements will be taken bilaterally and recorded in millimeters. The difference between the weighted and unweighted measurements will indicate foot posture: 5-9 millimeters is normal (neutral), 10 millimeters or more will indicate pronation (inward rotation), and 4 millimeters or less will indicate supination (outward rotation). This test is important for assessing the degree of pes planus.
Rotational Profile- Foot Progression Angle | Day 1
  The angle of foot progression is an important parameter to identify possible gait disorders and alignment problems by reflecting the rotational relationship between the femur, tibia and foot. For the test, two chairs facing each other will be placed 2 meters apart. The child will sit on a chair and the middle of the heel and the second toe will be marked with colored paint. The child will then stand up and walk naturally on a flat surface for about 5-6 steps towards the opposite chair and leave footprints. The child will then sit on the opposite chair and clean the paint from his feet. The footprints will be measured with a goniometer: one arm will be aligned with the direction of the footprints, the other will be parallel to the axis of the tibia. The angle between the foot and the tibia will be recorded in degrees.
Postural Control Assessment with the Biodex Balance System | Day 1
  Postural stability, limits of stability, and sensory integration of balance will be assessed using the Biodex Balance System®. It consists of a balance platform, arm supports, a screen, and a printer. The platform can be set to static or dynamic mode (12 levels; level 12 = most stable, level 1 = least stable with up to 20° movement in all directions). Prior to testing, children will be informed about the procedures. The heel and toe positions will be recorded based on medial-lateral (B-J), anterior, and posterior (1-21) axes. Arm support and screen height will be individually adjusted. Child-specific posture and identification data will be entered into the system. Three tests will be performed: postural stability, limits of stability, and sensory integration of balance.
Muscle Strength Assessment with Micro-FET 2 | Day 1
  Muscle tests will be performed using the MicroFET 2 digital hand dynamometer according to the device manual. The measurement will be performed in supine, prone, side-lying and sitting positions by preventing compensatory movements. During the test, the arms will be positioned so that they will not receive power from anywhere on/to the side of the body. Measurements will be performed bilaterally. While the child to whom the test is applied is expected to perform the requested movement with all his/her strength, the evaluating physiotherapist will apply resistance in the opposite direction in proportion to the strength. During the evaluation of the same muscle, a 30-second break will be given between repetitions, and a five-minute rest will be given before moving on to the test for a different muscle. Isometric muscle strength of the Iliopsoas, Gluteus Maximus, Gluteus Medius, Quadriceps, Hamstring, Tibialis Anterior, and Gastrosoleus muscles will be evaluated.
Functional Capacity Assessment with 6 Minute Walk Test | Day 1
  A 6 6-minute walk test will be done on a flat 30-meter track marked every 3 meters, with clear start and finish lines. Before the test, the child rests 15 minutes while contraindications will be checked. If none, blood pressure, oxygen saturation, pulse, and Borg scale scores for dyspnea and fatigue will be recorded. Medications taken will be noted. The child will be instructed to walk at their own pace for 6 minutes, allowed to stop or rest, and continue until "test is over" is announced. The test will start with "test is started" and end with "test is over." The timer runs continuously even if paused. The test ends if chest pain, severe breathlessness, cramps, unsteadiness, sweating, pallor, or oxygen saturation <85% occurs. Afterward, the child sits and post-test vitals and Borg scores will be recorded. Distance walked and any complaints during the test will be noted.
Lower Extremity Functional Scale | Day 1
  The Lower Extremity Functional Scale is a questionnaire that will evaluate the functional ability of the entire lower extremity in individuals with musculoskeletal disorders. This scale will question the difficulty experienced in various daily activities due to the problem in the lower extremity with 20 items. Each item is scored between 0-4 on a Likert scale (0=extremely difficult/too difficult to do the activity; 4=not difficult at all). The total score varies between 0-80 and the higher the score, the higher the functional level. A validity and reliability study has been conducted for the Turkish version of the scale to be used in evaluating lower extremity functions.

SECONDARY OUTCOMES:
Muscle Shortness/Flexibility- Thomas Test Measurement | Day 1
  The Thomas Test will be performed to evaluate shortness/tightness in the hip flexor muscle group, especially in the iliopsoas muscle. The child will be placed in the supine position, the lumbar spine will be fixed and the assessment will begin. During the test, while the assessed hip is in knee extension, the opposite hip and knee will be passively flexed by the physiotherapist, and the hip movement of the assessed side will be observed during this time. The Thomas test will be recorded as negative if no flexion movement is observed in the assessed hip. In the presence of shortness/tightness, the assessed hip is seen to be flexed, and in this case, the Thomas test will be recorded as positive.
Muscle Shortness/Flexibility- Popliteal Angle Measurement | Day 1
  The popliteal angle test will be used to evaluate shortness or tightness of the hamstring muscles. The hip and knee will be placed in a 90° flexion position while the child is in the supine position. While the physiotherapist passively moves the knee joint towards extension, the popliteal angle will be measured using a goniometer. While one arm of the goniometer is placed parallel to the lateral surface of the femur, the other arm is held parallel to the fibula head and the angle will be measured. The knee joint will be extended until it encounters resistance and the angle between the tibia and the vertical plane will be recorded as the popliteal angle.
Muscle Shortness/Flexibility- Silfverskiöld Test Measurement | Day 1
  Gastrocnemius assessment will be evaluated with the Silfverskiold test for all children participating in the study. The assessment will be performed bilaterally in supine positions where the child does not bear weight on their feet. The knee joint will be in full extension and 90° flexion, the subtalar joint will be in a neutral position, and the ankle dorsiflexion will be measured with the fixed arm of the universal goniometer on the fibula shaft and the mobile arm following the fifth metatarsal shaft. The measured angles will be recorded in degrees (°). Passive ankle dorsiflexion of ≤ 10° with the knee extended and a minimum of 10° increase in dorsiflexion with the knee flexed will be considered as isolated gastrocnemius muscle shortness.
Muscle Shortness/Flexibility- Ober Test Measurement | Day 1
  The Ober test will be an assessment to measure the length of the iliotibial band. During the test, the child will be placed in a supine position with the lower leg slightly flexed at the hip and knee. The upper leg will be in 90° flexion at the knee. Once positioning is complete, the physiotherapist will hold the ankle of the upper leg with one hand and stabilize the hip with the other hand. The leg will then be abducted and the knee extended and the leg moved until the femur is in line with the body. Finally, the thigh will be allowed to fall towards the surface in this plane and the result of the test will be judged by the amount of adduction of the hip. If the knee hangs in the air, the test will be recorded as positive; if the knee falls, the test will be recorded as negative.
Muscle Shortness/Flexibility- Duncal-Ely Test Measurement | Day 1
  The Duncan-Ely test will be used to evaluate the shortness and tightness of the rectus femoris muscle. While the child will be lying in the prone position, the hip will be fixed with one hand by the physiotherapist and the hip and knee will be kept in extension. In this position, the knee joint will be passively flexed to stretch the rectus femoris muscle on the tested side. If no shortness or tightness is observed in the rectus femoris muscle on the same side during the test and hip extension is maintained, the Duncan-Ely test will be recorded as negative. However, when the knee is flexed and a flexion movement is observed in the hip, the test will be recorded as positive.
Muscle Shortness/Flexibility- Sit-Reach Test Measurement | Day 1
  The sit-Reach test will be a frequently used test to evaluate the flexibility of the hamstring and lower back muscle groups. The S&R Sit and Reach® table will be used for this test. The child will sit in front of the table with dimensions of 55 cm long, 35 centimeters wide, and 30 centimeters high, and his/her feet will be positioned on the foot surface of the table. The child will be asked to place his/her hands on top of each other and stretch forward in a slow and controlled manner, bringing the ruler on the table forward. He/she will be asked to wait 1-2 seconds at the farthest point without stretching forward or backward. Scoring will be done according to the ruler on the table. (On this table, the child's ability to bring the ruler to the tips of his/her toes corresponds to 23 centimeters). The test will be repeated three times for each child to ensure reliability, and the highest value will be recorded in centimeters.
Pain Assessment with Visual Analog Scale | Day 1
  The Visual Analog Scale is a simple and reliable tool that is widely used to assess subjective experiences such as pain. It will consist of a 10-centimeter horizontal line with one end indicating "no pain" and the other end indicating "worst pain imaginable". Individuals will mark the point that reflects their perception of intensity, which will then be measured in millimeters or centimeters to obtain a numerical score. Higher values will indicate greater intensity. The Visual Analog Scale is valid and reliable in a variety of populations and conditions, including musculoskeletal pain.

OTHER OUTCOMES:
Demographic Information Form | Day 1
  Demographic data, including all children's gender, age, body weight, height and dominant side information, will be recorded before clinical evaluations. The body mass index (kilogram/meter2) of the child will be calculated and recorded with the recorded body weight (kilogram) and height (meter) values.
Leg Length Measurement | Day 1
  Leg Length Measurement, the child will be placed in a supine position. The legs will be positioned in extension and the muscles will be relaxed. The physiotherapist will measure and record the child's right leg length from the anterior superior iliac spine bone to the medial malleolus with a flexible metal tape measure. Measurements will be made bilaterally.
Ankle Joint Dorsiflexion Range of Motion Measurement | Day 1
  With the knee joint in full extension and 90° flexion, the subtalar joint in a neutral position, the ankle dorsiflexion will be measured with the fixed arm of the universal goniometer on the fibula shaft and the mobile arm following the fifth metatarsal shaft. The measured angles will be recorded in degrees (°). Measurements will be made bilaterally.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided